CLINICAL TRIAL: NCT06421454
Title: Clinical Trial for the Evaluation of Melatonin in the Treatment of Pressure Ulcers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Rioja Salud (Other)
Collaborators: Pharmamel S.L. (Industry); Universidad de Granada (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHM-2021-001
Record Dates: First submitted 2021-12-03; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Pressure Ulcer
Keywords: melatonin, ischemia
MeSH Terms: conditions — Pressure Ulcer; Ischemia | interventions — Melatonin; Hydrogels

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): Ulcers will be treated daily with melatonin cream for 8 weeks
  Interventions: Drug: Melatonin
- Control (Active Comparator): Ulcers will be treated daily with hydrogel for 8 weeks
  Interventions: Drug: Hydrogel

INTERVENTIONS:
Drug: Melatonin — Pressure Ulcer will be treated with a melatonin cream daily
  Other Names: Mel13Rx
  Arms: Melatonin
Drug: Hydrogel — Pressure ulcer will be treated with hydrogel daily as a comparator
  Other Names: Intransite
  Arms: Control

SUMMARY:
Melatonin has been shown to prevent cellular damage produced by oxidative stress or in situations of ischaemia, inhibiting the synthesis of oxidants and pro inflammatory factors such as pro-inflammatory cytokines, substances which are present in pressure ulcers and can affect the healing process, slowing it down. Melatonin gel has also been shown to prevent ulcers in the oral mucosa due to radiotherapy. Therefore, the hypothesis for this study is that the melatonin cream provides greater ulcer area reduction than standard pressure ulcer treatment.

DETAILED DESCRIPTION:
Melatonin has been shown to prevent cellular damage produced by oxidative stress or in situations of ischaemia, inhibiting the synthesis of oxidants and pro inflammatory factors such as pro-inflammatory cytokines, substances which are present in pressure ulcers and can affect the healing process, slowing it down. Melatonin gel has also been shown to prevent ulcers in the oral mucosa due to radiotherapy. Therefore, the hypothesis for this study is that the melatonin cream provides greater ulcer area reduction than standard pressure ulcer treatment.

In order to o determine the efficacy of melatonin in healing pressure ulcer it has been designed a multicentre, single-blind, randomized clinical trial comparing melatonin cream as an experimental pressure ulcer treatment versus control group with standard treatment based on moist environment wound healing with a time frame of 8 weeks. In order to assess the healing rate, changes in Resvech 2.0 scale scores will be measured, as well as the ulcer surface reduction. To avoid variability in measuring ulcer surface, it will be done by using software HELCOS after taking a photograph of the wound weekly. An intention-to-treat analysis will be carried out. The t-test or Mann-Whitney will be used to check difference of means in the reduction of the area of the ulcer and variation in the Resvech 2.0 scale. Survival curves will be used to check possible differences in the follow-up time until epithelization.

ELIGIBILITY:
Inclusion Criteria:

* Present at least one category II, III or IV pressure ulcer according to National Group for the Study and Assessment of Pressure Ulcers (GNEAUPP) classification.
* Ulcer area between 1 and 100 cm2.
* People over 18 years of age who have freely given their informed consent in writing of their own volition or it has been given on their behalf by a legal guardian

Exclusion Criteria:

* Ulcer of category I, non-classifiable or affecting internal tissues, but with no break in the skin
* People currently undergoing chemotherapy treatment or who have done so in the previous 6 months
* People with a presumed life expectancy of less than 6 months or in palliative care.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Epithelialisation | Up to 8 weeks
  Percentage of completely epithelialized ulcers

SECONDARY OUTCOMES:
Pressure ulcer area | Up to 8 weeks
  Percentage of reduction in pressure ulcer area

CONTACTS AND LOCATIONS:
Overall Officials: Marco Aldonza -Torres, Principal Investigator — Fundacion Rioja Salud

IPD SHARING:
Plan to Share IPD: No